CLINICAL TRIAL: NCT05891964
Title: Outcome of Treatment With Secukinumab in the Treatment of Moderate to Severe Plaque Psoriasis at Tertiary Care Hospital.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jinnah Postgraduate Medical Centre (Other Government)
Responsible Party: Principal Investigator, Faiza Inam Siddiqui, Principal Investigator, Jinnah Postgraduate Medical Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NO.F2-81/2022-GENL/252/JPMC
Record Dates: First submitted 2023-03-22; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Plaque Psoriasis
Keywords: Plaque Psoriasis; Secukinumab Injection; Outcome
MeSH Terms: interventions — secukinumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Secukinumab (Experimental): Injection Secukinumab 150mg subcutaneously will be administered at weeks 0, 1, 2, 3, 4, and then monthly for 5 months.
  Interventions: Drug: Secukinumab Injection

INTERVENTIONS:
Drug: Secukinumab Injection — Injection Secukinumab 150mg subcutaneously will be administered at weeks 0, 1, 2, 3, 4, and then monthly for 5 months.
  Other Names: Cosentyx

SUMMARY:
Psoriasis is one of the most common immune-mediated inflammatory disorders characterized by a chronic course. It affects approximately 2-3% of the world's population Psoriasis may be provoked by environmental factors in patients with genetic predispositions. Psoriasis is phenotypically characterized by thickened, red, scaly plaques and systemic inflammation, it is also associated with multiple comorbidities, such as cardiovascular disease, stroke, hypertension, metabolic diseases, chronic kidney disease, and joint destruction. Psoriasis is pathogenically driven by proinflammatory cytokines and mediated by T and dendritic cells. Inflammatory myeloid dendritic cells release interleukin (IL) 23 and IL-12 to activate IL-17-producing T cells, Th1 cells, and Th22 cells to produce psoriatic cytokines like IL-17, interferon (IFN) γ, TNF, and IL-22. These cytokines mediate the effects on keratinocytes. Secukinumab is a recombinant human monoclonal antibody that specifically binds to a proinflammatory cytokine released by T-helper-17 (Th17) cells, IL-17A. It blocks its binding with IL-17R and the expression of cytokines. This blockade normalizes the inflammatory processes and combats epidermal hyperproliferation, T-cell infiltration, and exaggerated expression of pathogenic genes.

DETAILED DESCRIPTION:
Plaque psoriasis is a chronic autoimmune skin disorder characterized by the formation of thick, scaly plaques on the skin surface. It affects millions of individuals worldwide and significantly impacts their quality of life. While several treatment options exist, a substantial number of patients with moderate to severe plaque psoriasis fail to achieve satisfactory results or experience intolerable side effects with conventional therapies.

Psoriasis is pathogenically driven by proinflammatory cytokines and mediated by T cells and dendritic cells. In recent years, the advent of biologic agents targeting specific immune pathways has revolutionized the management of psoriasis. Secukinumab, a fully human monoclonal antibody that selectively inhibits interleukin-17A, has shown promising results in randomized controlled trials and real-world studies. However, there remains a need to assess the real-world effectiveness and safety of Secukinumab in routine clinical practice, particularly in patients with moderate to severe plaque psoriasis who may have diverse characteristics and treatment histories.

This observational study aims to evaluate the real-world effectiveness and safety of Secukinumab in patients with moderate to severe plaque psoriasis. By collecting data from a diverse patient population in routine clinical settings, we aim to provide valuable insights into the outcomes and experiences of patients receiving Secukinumab outside the controlled environment of clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Known plaque psoriasis
* Either gender
* Age 30-80 years.

Exclusion Criteria:

* Patients with history of eczema.
* Patients with history connective tissue disorder, vasculitis malignancy, seropositive or seronegative arthritis.
* Patients with history of malignancy.
* Patient with history of hepatis B, C or AIDS.
* Immunocompromised patients.
* Pregnant patients assessed by history and confirmed by dating scan.
* Patients with history of chronic liver disease, chronic kidney disease, asthma, acute coronary syndrome, congestive heart failure and chronic obstructive pulmonary disease will be excluded.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-06-05 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of Secukinumab in the treatment of moderate to severe plaque psoriasis | From day of randomisation until final dose of drug,assessed upto 12 months.
  Efficacy will be assessed using psoriasis area and severity index. The minimum score of psoriasis area and severity index is 0 and the maximum score is 72. All patients who will be presented with 75% reduction in the Psoriasis Area and Severity Index at the end of the therapy compared to baseline will be labelled as positive for efficacy.

SECONDARY OUTCOMES:
Mean difference of Psoriasis Area and Severity Index score before and after the treatment | From day of randomisation until final dose of drug,assessed upto 12 months.
  Psoriasis area and severity index score difference before the treatment and after the treatment will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Faiza I Siddiqui, Principal Investigator — Jinnah post graduate Medical centre; Rabia Ghafoor, Principal Investigator — Jinnah post graduate Medical centre
Locations (1):
- Jinnah Post graduate Medical centre, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No